CLINICAL TRIAL: NCT06872190
Title: Using Clinical Decision Support to Provide Social Risk-Informed Care for Opioid Use Disorder in the Emergency Department
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: Single | Purpose: Health Services Research
Other Study IDs: 24-41722; K23DA060993 (NIH)
Record Dates: First submitted 2025-03-06; First posted 2025-03-12 (Actual); Last update posted 2025-05-07 (Actual); Status verified 2025-05

CONDITIONS: Opioid Use Disorder; Social Determinants of Health (SDOH)
Keywords: social risk-informed care; clinical decision support; opioid use disorder
MeSH Terms: conditions — Opioid-Related Disorders

STUDY DESIGN:
Intervention Model Description: The investigators will first deploy CDSv1 and collect outcomes with CDSv1, while they build CDSv2. After a brief wash-in period, they will deploy CDSv2 and collection outcomes on CDSv2.
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ED-Based Clinical Decision Support for Opioid Use Disorder (Active Comparator): Emergency providers will have access to the basic ED-based clinical decision support tool for opioid use disorder.
  Interventions: Other: ED-Based Clinical Decision Support for Opioid Use Disorder
- Social Care-Enhanced Clinical Decision Support for Opioid Use Disorder (Experimental): Emergency providers will no longer have access to the basic ED-based clinical decision support tool for opioid use disorder, but will instead have access to the social care-enhanced clinical decision support tool for opioid use disorder.
  Interventions: Other: Social Care-Enhanced Clinical Decision Support for Opioid Use Disorder

INTERVENTIONS:
Other: ED-Based Clinical Decision Support for Opioid Use Disorder — The original clinical decision support (CDS) tool, EMergency department initiated BuprenorphinE for opioid use Disorder or EMBED, was designed by researchers at Yale to support emergency department (ED) clinicians with varying levels of experience prescribing buprenorphine for patients with opioid use disorder (OUD). The tool alerts ED providers of a patient who is potentially eligible for MOUD using Epic's storyboard. The provider must then click on the notification to open the OUD evaluation tool, which has multiple components: OUD assessment, OUD diagnosis, withdrawal assessment, and readiness for treatment. These components are then paired with an orderset, "ED Opioid Use Disorder Treatment" that includes nursing orders, prescriptions for buprenorphine and ancillary medications, and substance use disorder discharge resources.
  Other Names: CDSv1
  Arms: ED-Based Clinical Decision Support for Opioid Use Disorder
Other: Social Care-Enhanced Clinical Decision Support for Opioid Use Disorder — The investigators will use human-centered design to adapt the basic CDS tool to incorporate patient social needs, involving patients, staff, and end-user ED clinicians in the iterative design process. This tool is being actively developed.
  Other Names: CDSv2
  Arms: Social Care-Enhanced Clinical Decision Support for Opioid Use Disorder

SUMMARY:
The overarching goal of this proposal is to integrate patient social risk information into an existing electronic health record (EHR)-based clinical decision support (CDS) tool (CDSv1) to facilitate emergency department (ED)-initiated, social risk-informed opioid use disorder (OUD) medication treatment and ultimately improve treatment adherence and follow up. The investigators will evaluate the feasibility and acceptability of the social care-enhanced CDS tool, CDSv2, (compared to CDSv1) at a single study site (UCSF) as an intervention to increase medication treatment adherence and follow up for adult ED patients experiencing opioid use disorder using a mixed-methods, before-after approach.

DETAILED DESCRIPTION:
Over 2.7 million people suffer from opioid use disorder (OUD) in the United States (US), resulting in more than 80,000 opioid overdose deaths in 2021. Medications for opioid use disorder are underused disproportionately in patients living in poverty, whose unmet food, housing, and transportation needs impede access to medications and routine healthcare. Emergency departments (EDs) are the primary (and often only) healthcare access points for vulnerable populations with social needs, including people with OUD. In response, healthcare professional organizations have increasingly called for ED-initiated medications for OUD (MOUD), which has been shown to lead to better adherence compared to referrals to treatment alone.

Clinical decision support (CDS) tools in electronic health records (EHRs) can be used to support ED-initiated MOUD. They enhance care quality by providing actionable information to clinicians in real time; a study of a CDS tool for MOUD showed that it significantly increased the number of MOUD prescribers. A major risk of ED-initiated MOUD, however, is that it could lead to inequitable outcomes unless closely paired with efforts to connect patients to services that also address social needs. For instance, patients with food or housing insecurity are unlikely to prioritize adherence to MOUD over meeting their basic material needs; patients with MOUD who lack reliable transportation may be unable to access follow up care for MOUD. Linking social interventions to MOUD initiation may improve the likelihood of adherence to treatment and follow-up care. Though CDS tools that use patients' social risk data have been developed to improve care for other chronic diseases, e.g., hypertension and diabetes, to date, the CDS tools that facilitate ED-initiated MOUD have not been designed to harness social risk information to improve MOUD care planning. There is an urgent need to design and test a CDS tool that simultaneously facilitates MOUD initiation and helps identify and intervene on patients' social needs.

The overarching goal of this project is to evaluate the feasibility and acceptability of a social care-enhanced CDS tool (CDSv2) designed to facilitate ED-based, social risk-informed MOUD compared to an existing CDS tool for ED-based MOUD (CDSv1), with the ultimate goal of improving treatment adherence and follow up for ED patients experiencing OUD.

Specific Aim: Assess the feasibility and acceptability of the social care-enhanced CDS tool (CDSv2, compared to CDSv1) at the UCSF ED as an intervention to improve medication treatment adherence and follow up for adult ED patients experiencing OUD. The investigators will perform a mixed-methods, before-after pilot study evaluating the basic CDS tool (CDSv1) and the social care-enhanced CDS tool (CDSv2) over 28 months. To assess feasibility of patient recruitment and primary endpoint collection (e.g, adherence, follow up), the investigators will perform chart review and outreach to patients. To measure clinician utilization and acceptability, the investigators will collect EHR-based audit log and survey data. The investigators will also conduct semi-structured interviews with a purposive sample of ED clinicians and patients to further capture their experiences (acceptability) with the social care-enhanced CDS tool and the basic CDS tool.

The expected sample size of 300 will include 240 providers and 60 patients.

ELIGIBILITY:
Inclusion criteria:

* All University of California, San Francisco ED providers (residents, attendings, advanced practice providers) who have used either CDSv1 or CDSv2 will be eligible to participate in surveys and interviews regarding feasibility and acceptability.
* English-speaking patients ≥18 years of age presenting to the UCSF ED with opioid use disorder who receive medication treatment (as a result of CDSv1 or CDSv2) will be eligible to participate.

Exclusion criteria:

- Participants will be excluded if:

* they have a medical or psychiatric condition requiring hospitalization at the index ED visit,
* are actively suicidal, are cognitively impaired,
* present from an extended care facility, or
* require opioids for a pain condition.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2025-04-20 (Actual); Primary Completion 2027-07 (Estimated); Study Completion 2027-07 (Estimated)

PRIMARY OUTCOMES:
CDSv1 clinician launch | 12 months
  Percentage of ED clinicians who launch CDSv1 for patients with OUD
CDSv1 encounter launch | 12 months
  Percentage of eligible encounters (i.e., encounters including patients with OUD as defined by the EHR-derived phenotype) where CDSv1 was launched by clinician
CDSv2 clinician launch | 12 months
  Percentage of ED clinicians who launch CDSv2 for patients with OUD
CDSv2 encounter launch | 12 months
  Percentage of eligible encounters (i.e., encounters including patients with OUD as defined by the EHR-derived phenotype) where CDSv2 was launched by clinician
CDSv1 adherence to OUD treatment recommendations | 12 months
  For ED visits in which CDSv1 is launched, investigators will assess the percentage of times either buprenorphine, methadone, or naltrexone was prescribed by an ED clinician
CDSv2 adherence to OUD treatment recommendations | 12 months
  For ED visits in which CDSv2 is launched, investigators will assess the percentage of times either buprenorphine, methadone, or naltrexone was prescribed by an ED clinician
CDSv2 adherence to social care recommendations | 12 months
  For ED visits in which CDSv2 is launched, investigators will assess the percentage of times social care recommendations (to be determined, based on results from Aim 2) were followed by ED clinicians
CDSv1 acceptability | During first 6 months of CDSv1 deployment
  Acceptability of Intervention Measure 4-item survey to assess clinician acceptability of CDSv1. Response scales range from "1 = Completely disagree" to "5 = Completely agree", with higher scores indicating greater success.
CDSv1 appropriateness | During first 6 months of CDSv1 deployment
  Intervention Appropriateness Measure 4-item survey to assess clinician perception of CDSv1 appropriateness. Response scales range from "1 = Completely disagree" to "5 = Completely agree", with higher scores indicating greater success.
CDSv2 acceptability | During first 6 months of CDSv2 deployment
  Acceptability of Intervention Measure 4-item survey to assess clinician acceptability of CDSv2. Response scales range from "1 = Completely disagree" to "5 = Completely agree", with higher scores indicating greater success.
CDSv2 appropriateness | During first 6 months of CDSv2 deployment
  Intervention Appropriateness Measure 4-item survey to assess clinician perception of CDSv2 appropriateness. Response scales range from "1 = Completely disagree" to "5 = Completely agree", with higher scores indicating greater success.
Patient recruitment CDSv1 | 12 months
  Number of patients who receive OUD medication as a result of CDSv1 who are enrolled for primary outcome ascertainment
Patient recruitment CDSv2 | 12 months
  Number of patients who receive OUD medication as a result of CDSv2 who are enrolled for primary outcome ascertainment
ED clinicians' perceptions of CDSv1 | Within first 8 months of CDSv1 deployment
  Themes emerging from semi-structured qualitative interviews exploring clinician perceptions of CDSv1
ED patients' perceptions of CDSv1 | Within first 8 months of CDSv1 deployment
  Themes emerging from semi-structured qualitative interviews exploring patient perceptions of receiving treatment from CDSv1
ED clinicians' perceptions of CDSv2 | Within first 8 months of CDSv2 deployment
  Themes emerging from semi-structured qualitative interviews exploring clinician perceptions of CDSv2
ED patients' perceptions of CDSv2 | Within first 8 months of CDSv2 deployment
  Themes emerging from semi-structured qualitative interviews exploring patient perceptions of receiving social risk-informed treatment from CDSv2
Feasibility of primary endpoint collection for CDSv1 | 13 months
  Percentage of participants for whom data on OUD medication adherence and follow up are successfully collected at 30 days for CDSv1
Feasibility of primary endpoint collection for CDSv2 | 13 months
  Percentage of participants for whom data on OUD medication adherence and follow up are successfully collected at 30 days for CDSv2

SECONDARY OUTCOMES:
CDSv1 treatment adherence | 13 months
  Proportion of participants adherent to the same OUD medication prescribed using CDSv1 at 30 days post-ED visit
CDSv1 follow up | 13 months
  Proportion of participants receiving formal inpatient, outpatient, or ED-based addiction treatment services at 30 days post-ED visit for CDSv1
CDSv2 treatment adherence | 13 months
  Proportion of participants adherent to the same OUD medication prescribed using CDSv2 at 30 days post-ED visit
CDSv2 follow up | 13 months
  Proportion of participants receiving formal inpatient, outpatient, or ED-based addiction treatment services at 30 days post-ED visit for CDSv2

CONTACTS AND LOCATIONS:
Overall Officials: Melanie F Molina, MD, MAS, Principal Investigator — University of California, San Francisco
Locations (1):
- University of California, San Francisco, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: No